CLINICAL TRIAL: NCT05783427
Title: An Evaluation of a Liberal Hydration Regimen Before Elective Caesarean Section Using
Brief Title: An Evaluation of a Liberal Hydration Regimen Before Elective Caesarean Section Using Beside Gastric Ultrasound
Status: Completed | Type: Observational
Sponsor: Coombe Women and Infants University Hospital (Other)
Responsible Party: Principal Investigator, Ryan Howle, Principal Investigator, Consultant Anaesthesiologist, Coombe Women and Infants University Hospital
Other Study IDs: GUS123
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Aspiration; Gastric Contents, Anesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: liberal hydration — evaluate the effect of 'Sip Til Send' on overall gastric volume pregnant women undergoing elective caesarean delivery
  Other Names: 'sip til send'

SUMMARY:
The aim of this study is to compare the residual gastric volumes in non-labouring parturients prior to elective Caesarean delivery when fully fasted as per European Society of Anaesthesia pre-operative fasting guidelines against the 'Sip Til Send' fasting guideline via a paired cohort study. The primary hypothesis is that 'Sip Til Send' would be non-inferior to standard fasting at minimising the residual gastric volume prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* planned caesarean delivery under regional anaesthesia
* adhered to national fasting guidance of 6 hrs for food and 2 hours for clear fluids

Exclusion Criteria:

* age less than 18
* inability to understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women who are undergoing a planned elective caesarean delivery
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
gastric volume | 3 months
  whether a liberal hydration protocol can be safely provided to pregnant women undergoing elective caesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Howle, Principal Investigator — Coombe Womens Hospital
Locations (1):
- Coombe Women's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harnett C, Connors J, Kelly S, Tan T, Howle R. Evaluation of the 'Sip Til Send' regimen before elective caesarean delivery using bedside gastric ultrasound: A paired cohort pragmatic study. Eur J Anaesthesiol. 2024 Feb 1;41(2):129-135. doi: 10.1097/EJA.0000000000001926. Epub 2023 Nov 20. PMID 37982593